CLINICAL TRIAL: NCT06815770
Title: Efficacy and Safety of Continuous Infusion of Terlipressin vs Bolus Terlipressin in ACLF Patients With Acute Esophageal Variceal Bleed: Pilot Study
Brief Title: Efficacy and Safety of Continuous Infusion of Terlipressin vs Bolus Terlipressin in ACLF Patients With Acute Esophageal Variceal Bleed
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-22
Record Dates: First submitted 2025-01-30; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus terlipressin (Active Comparator): 2 mg initially every 4 hourly for 2 days and then 1 mg every 4 hrs.
  Interventions: Drug: Terlipressin Injectable Product
- Continous Infusion of Terlipressin (Experimental): Administered as a continuous infusion at 4 mg/24 hours. After 12 hours, if the hepatic venous pressure gradient (HVPG) does not show a reduction of less than 10%, increase the dose to 6 mg/24 hours.
  Interventions: Drug: Terlipressin Injectable Product

INTERVENTIONS:
Drug: Terlipressin Injectable Product — Terlipressin Injectable Product

SUMMARY:
Acute portal hypertension, as measured by rapid rise in hepatic venous pressure gradient (HVPG) can lead to further dreaded complications, including acute variceal bleeding (AVB) AVB: 6-week mortality rates of around 15-20% in patients with chronic liver disease without ACLF.The overall prevalence of UGH in cirrhotic patients with AD was 34.4% and 35.7% in patients with ACLF.AVB is a well-recognized precipitant leading to the occurrence and development of ACLF. AVB is a well-recognized precipitant leading to the occurrence and development of ACLF. Medical therapy for esophageal variceal bleeding (EVB) aims to reduce the splanchnic blood flow and portal pressure. The most common vasoactive agents include terlipressin, vasopressin, somatostatin, and octreotide.

DETAILED DESCRIPTION:
Aim and Objective - To assess the safety and efficacy of continuous terlipressin vs. Bolus terlipressin in the management of acute esophageal variceal bleeding in ACLF.

Study population: Adult patients (age ≥ 18 years) diagnosed with ACLF presenting with upper GI bleeding due to esophageal varices Study design: Pilot study Study period: 1 year Sample size: 60

Intervention:

Group I- Intravenous terlipressin (administered as a continuous infusion at 4 mg/24 hours). After 12 hours, if the hepatic venous pressure gradient (HVPG) does not show a reduction of less than 10%, increase the dose to 6 mg/24 hours.

Group II- Intravenous terlipressin (2 mg initially every 4 hourly for 2 days and then 1 mg every 4 hrs)

Monitoring and assessment: All patients would undergo vital and baseline parameter screening before randomization. Based on randomization they will receive either steroid or plasma exchange followed by steroid

Adverse effects:

Acute Diarrhea, chest pain, Arterial hypertension, Cardiac arrhythmias, Acute abdomen Stopping rule: chest pain, alteration of ECG, cyanosis, bradycardia, severe allergic rashes

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age ≥ 18 years) diagnosed with ACLF presenting with due to esophageal varices bleeding.

Exclusion Criteria:

1. Age < 18 years
2. History of coronary heart disease or ventricular arrhythmia,
3. Stroke or transient ischemic attack,
4. Bronchial asthma,
5. Epilepsy,
6. Pregnancy,
7. Rebleeding.
8. HCC
9. Gastric variceal bleed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Hepatic venous Pressure Gradient (HVPG) reduction of more than 10% from baseline at 12-24 hours in both arms. | 12-24 hours

SECONDARY OUTCOMES:
Failure to control hemostasis | 5 days
Terlipressin-related complications within 5 days i.e. safety of the drug | 5 days
Number of blood transfusions at 5 days | 5 days
Rebleed within 42 day | 42 days
Incidence of post-bleed Acute Kidney Injury within 5 days | 5 days
6 weeks mortality in both groups. | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided